CLINICAL TRIAL: NCT06763471
Title: Single Unit Neurophysiological Architecture of the Neocortex (SUNAN)
Brief Title: Measuring Single Neuron Activity in the Brain
Acronym: SUNAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Francis Crick Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 159671
Record Dates: First submitted 2024-12-20; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Neurological Diseases or Conditions
Keywords: Neuron activity; Single unit; Neurosurgery; Neuropixels; Neurophysiology; Cortical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neuropixels recording (Experimental): Participants undergoing planned neurosurgery that undergo a maximum of 15 minutes neurophysiological recording using Neuropixels
  Interventions: Device: Neuropixels recording intraoperatively during planned neurosurgery

INTERVENTIONS:
Device: Neuropixels recording intraoperatively during planned neurosurgery — The SUNAN study is a basic science study involving a procedure to record single-unit neurophysiological activity with human participants who are already undergoing a transcranial neurosurgical procedure on the brain.
  As part of the surgery, a region of cerebral cortex on the convexity of the brain will be:
  * Resected e.g., as removal of part of a tumour or epilepsy focused. Or
  * Transgressed as part of the surgical approach to reach a deeper target e.g., resection of a deep tumour or cavernoma.
  Or
  • Transgressed by the passage of a surgical implant e.g., a ventriculoperitoneal shunt catheter or deep brain stimulation electrode.
  Within this region of the brain that is going to be resected or transgressed, the research team will undertake a single-unit resolution neurophysiological recording (NR) using a digital neural probe (Neuropixels) for a maximum of 15 minutes.

SUMMARY:
The SUNAN (Single Unit Neurophysiological Architecture of the Neocortex) study aims to understand how individual brain cells called neurons interact and communicate, and how the neurons can be affected in neurological disease. Using an advanced digital probe called the "Neuropixels probe," which is as thin as a human hair, the investigators can record electrical activity from individual neurons on the outmost layer of the brain (cerebral cortex). This electrical (neurophysiological) activity recording technique allows the investigators to isolate and monitor single-neuron activity from the human brain during planned neurosurgical operations in real time.

DETAILED DESCRIPTION:
The SUNAN study plans to recruit fifty patients scheduled for brain surgery, such as for tumour removal or operations that involve the fluid (cerebrospinal fluid) within the brain, at the National Hospital for Neurology and Neurosurgery. Participation is voluntary, and the suitability will be assessed by the participant's neurosurgeon.

Patients who participate in SUNAN will undergo their planned neurosurgery as per standard of care with the additional step of a neurophysiological recording made from the brain using a Neuropixels probe. This recording step and the data collected will not affect the rest of the patients care which will proceed in the usual way and the data is collected solely for scientific purposes.

The investigators believe that the insights gained from these electrical recordings from individual neurons will deepen our understanding of brain function and potentially lead to improved diagnosis and treatment of neurological diseases.

ELIGIBILITY:
1. Aged 18 years and over.
2. Documented informed consent to participate.
3. Undergoing a transcranial neurosurgical procedure at the National Hospital for Neurology and Neurosurgery (NHNN) in which part of the cerebral cortex will be:

   * Resected e.g., as removal of part of a tumour or epilepsy focused. Or
   * Transgressed as part of the surgical approach to reach a deeper target e.g., resection of a deep tumour or cavernoma.

   Or

   • Transgressed by the passage of a surgical implant e.g., a ventriculoperitoneal shunt catheter or deep brain stimulation electrode.
4. Surgery felt to be technically suitable for the neurophysiological recording technique by the Chief Investigator and responsible Consultant Neurosurgeon. For example, participants having surgery in an unusual position may present problems for the neurophysiological recording step.

Exclusion Criteria:

1. Participants who lack the capacity to give informed consent.
2. Participants who are pregnant or breast feeding at the time of surgery.
3. Participants deemed to be unsuitable for recruitment to the study by the responsible Consultant Neurosurgeon. If in the view of the treating consultant involvement in the study would compromise the patient's surgery or present an unacceptable risk to them, they will not be recruited to the study. For example, if the participant does not meet the standard of care preoperative checks.
4. Concern from the Consultant Neurosurgeon or treating Anaesthetist that there would be an unreasonable burden on the patient to participate in the study. For example, risk due to increased length of anaesthetic time.
5. For participants requiring anaesthesia for their pre-planned brain surgery, an American Society of Anaesthesiologists (ASA) physical status classification system score of 4 and higher.
6. Participants unable to understand English sufficiently well to read the patient facing documents and consent in English.
7. Participants not undergoing their treatment through National Health Service (NHS) care (i.e. private patients are excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Single units isolated | Timepoint - At time of planned neurosurgery.
  Outcome name - Descriptive reporting on the number of well isolated single neuronal units observed during neurophysiological recording of the brain during planned neurosurgery.
  Metric/method of measurement - Neurophysiological activity of the brain will be described through analysis of electrical activity recorded. The detection of spikes represents depolarisation of single neuronal units ("single-units"). Well isolated single-units will be defined by clustering metrics, interval spike interval violations and/or other neurophysiological analysis. Descriptive reporting will include the number of individual units recorded, their spiking rates and correlation.

SECONDARY OUTCOMES:
Experience of using large scale single-unit recording | Through study completion, an average of 1 year
  Secondary outcome measures will be reported for each participant to gather information on the recording technique. For example, a description of the recording setting may include the arrangement of ground and reference electrodes as well as the operative set-up.
  Reporting on the experience of using large scale single-unit recording techniques in humans undergoing neurosurgery.
Iterations made to the surgical and electrophysiological technique | Through study completion, an average of 1 year
  Reporting on iterations made to the surgical and electrophysiological technique over the course of the study.
Potential refinements in technique | Through study completion, an average of 1 year
  Reporting on potential refinements that could be made to the described technique which could enable better quality data and that could be of benefit to other researchers conducting similar work. For example, equipment set-up/noise restrictions in theatre.

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plans for the current study are unknown and will be made available at a later date.